CLINICAL TRIAL: NCT03205813
Title: Prospective Study of Pain After Spinal Morphine for Cesarean Section and Analysis of Factors Involved in Moderate to Severe Pain
Brief Title: Prospective Study of Pain After Spinal Morphine for Cesarean Section and Factors Involved in Moderate to Severe Pain
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 164/2560(EC2)
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Pain, Postoperative
Keywords: Pain, Postoperative; Cesarean delivery; Intrathecal morphine
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spinal block with intrathecal morphine is a popular anesthetic technique in cesarean delivery. This technique brings about good maternal and neonatal outcomes as well as provides good postoperative pain control. Systematic review showed intrathecal morphine produced long period of pain control up to 27 hours. However, some patients still experienced moderate to severe pain which defined as postoperative pain score >,= 4. From our institute survey, there were more than 50 percents of patients undergoing cesarean delivery receiving spinal block with intrathecal morphine experienced moderate to severe pain in the first 24 hours.

The aim of the study is to determine the actual incidence and associated factors of patients whom experienced moderate to severe pain after spinal anesthesia with intrathecal morphine 200 mcg in cesarean delivery.

DETAILED DESCRIPTION:
Spinal block with intrathecal morphine is a popular anesthetic technique in cesarean delivery. This technique brings about good maternal and neonatal outcomes as well as provides good postoperative pain control. Systematic review showed intrathecal morphine produced long period of pain control up to 27 hours. However, some patients still experienced moderate to severe pain which defined as postoperative pain score >,= 4. From our institute survey, there were more than 50 percents of patients undergoing cesarean delivery receiving spinal block with intrathecal morphine experienced moderate to severe pain in the first 24 hours. Failure in achieve adequate pain control results in poor maternal satisfaction, effect breast feeding and may lead to chronic wound pain.

The aim of the study is to determine the actual incidence of patients whom experienced moderate to severe pain after spinal anesthesia with intrathecal morphine 200 mcg in cesarean delivery. Also, factors that may involved moderate to severe postoperative pain will be analyzed and reported.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Elective cesarean section
* Patient accept spinal anesthesia
* ASA classification I-II
* Understand numerical rating scale for pain score

Exclusion Criteria:

* Not understand Thai
* Contraindicated in spinal anesthesia with intrathecal morphine
* Complicated pregnancy that general anesthesia may required for cesarean delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Patients undergoing elective cesarean delivery
Sampling Method: Non-Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of moderate to severe pain | The first 24 hours postoperatively
  Incidence of moderate to severe pain, pain score >,= 4

SECONDARY OUTCOMES:
Factors associated with moderate to severe pain | The first 24 hours postoperatively
  Factors associated with moderate to severe pain, pain score >,= 4
Incidence of moderate to severe pain in the 2nd postoperative day | Form 24 hours to 48 hours postoperatively
  Incidence of moderate to severe pain (pain score >,= 4) in the 2nd postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Patchareya Nivatpumin, M.D., Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Bangkok, Thailand
Locations (1):
- Anesthesiology department, Siriraj hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nivatpumin P, Pangthipampai P, Dej-Arkom S, Aroonpruksakul S, Lertbunnaphong T, Ngam-Ek-Eu T. Gestational diabetes and intraoperative tubal sterilization are risk factors for high incidence of pain after cesarean delivery: a prospective observational study. Ann Palliat Med. 2022 Apr;11(4):1170-1178. doi: 10.21037/apm-21-2139. Epub 2021 Dec 17. PMID 34930012